CLINICAL TRIAL: NCT07405515
Title: Pathophysiology of Dysautonomia and Postural Tachycardia Syndrome (POTS) in Post-viral Syndromes and COVID-19
Acronym: fBRI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: FBRI LLC (F-Prime Capital) (Unknown)
Responsible Party: Principal Investigator, Peter Novak, MD, PhD, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P000633; 2022A018462 (Other Grant/Funding Number: FBRI LLC [Industry])
Record Dates: First submitted 2026-01-30; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: POTS; POTS - Postural Orthostatic Tachycardia Syndrome; Dysautonomia; Autonomic Dysfunction
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases; Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Dysautonomia/POTS (Experimental): Participants with a diagnosis of dysautonomia or POTS will undergo a single blood draw of approximately 30 mL for research purposes, including immune system and genetic analyses. Samples will be coded and stored for future research. No therapeutic intervention is administered.
  Interventions: Other: Blood Sample Collection
- Healthy Control Participants (Experimental): Healthy volunteers without dysautonomia or POTS will undergo the same single blood draw of approximately 30 mL for research purposes, including immune system and genetic analyses. Samples will be coded and stored for future research. No therapeutic intervention is administered.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — All participants, including people diagnosed with dysautonomia/POTS and healthy control participants, will undergo a single blood draw of approximately 30 mL (about 2 tablespoons). The blood will be collected for research purposes, including immune system and genetic analyses, and stored in a coded fashion for future research. No therapeutic intervention, drug, or device will be administered.

SUMMARY:
This study aims to better understand the biological mechanisms underlying dysautonomia and postural orthostatic tachycardia syndrome (POTS), including how these conditions may be related to COVID-19. Participants will attend a single research visit lasting approximately one hour, during which a blood sample will be collected for immune system and genetic analyses. Information from participants' medical records may also be reviewed to support the research. The knowledge gained from this study may help improve understanding, diagnosis, and treatment of dysautonomia in the future.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged ≥18 years
* Diagnosis of idiopathic POTS (neuropathic form with evidence of neurodegeneration on skin biopsy) or Long COVID with or without POTS
* Age-matched healthy controls with normal autonomic testing
* Symptoms consistent with POTS: orthostatic intolerance ≥3 months with a clearly defined antecedent event (infection, travel, surgery)
* Orthostatic tachycardia >30 BPM without orthostatic hypotension, associated with reduced cerebral orthostatic blood flow and hypocapnia
* Availability of electronic health record

Exclusion Criteria:

* Known causes of small fiber neuropathy, including: diabetes, amyloidosis, lupus, Sjogren syndrome, cancer, Ehlers-Danlos syndrome
* Other medical explanations for POTS symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune system profiling of peripheral blood: cytokines, immune cell populations, and inflammatory mediators | Single research visit per participant; outcomes assessed at the time of sample collection and analysis. Starting from 2024 and expected to end in 2027.
  Peripheral blood will be collected from participants with POTS/dysautonomia, Long COVID, and healthy controls during a single research visit (~1 hour). Samples will be analyzed to quantify cytokines, immune cell subsets, and inflammatory mediators to identify immune signatures associated with dysautonomia and PASC. Data will be aggregated by participant group and analyzed for differences in immune profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data due to privacy concerns and the sensitive nature of genetic and immune system information. Data will be de-identified and stored securely, and only aggregate results will be shared in publications.